CLINICAL TRIAL: NCT05093413
Title: Olfactory Decision-making and Deprived Sleep
Acronym: ODDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Christina Zelano, Principal Investigator, Northwestern University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: STU00215342
Record Dates: First submitted 2021-09-29; First posted 2021-10-26 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Sleep Deprivation
MeSH Terms: conditions — Sleep Deprivation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fully slept first; Sleep deprived second (Experimental): Participants will be fully slept during the first experimental visit and sleep deprived during the second experimental visit
  Interventions: Behavioral: Sleep deprivation
- Sleep deprived first; Fully slept second (Experimental): Participants will be sleep deprived during the first experimental visit and fully slept during the second experimental visit
  Interventions: Behavioral: Sleep deprivation

INTERVENTIONS:
Behavioral: Sleep deprivation — Fully slept: Sleep habitual amount (i.e., go to sleep at habitual bedtime and wake up at habitual wake time) Sleep deprived: Reduce sleep by 50% (i.e., go to sleep at habitual bedtime and wake up early)

SUMMARY:
This research study will use magnetic resonance imaging (MRI) and olfactory stimuli to better understand the connection between sleep deprivation, brain activity, and olfaction in humans.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Fluent English speakers

Exclusion Criteria:

* History of neurological conditions (e.g., epilepsy, dementia, multiple sclerosis, brain tumors, etc.)
* History of psychiatric conditions (e.g., general anxiety disorder, depression, schizophrenia, obsessive-compulsive disorder, post-traumatic stress disorder, attention deficit hyperactivity disorder, alcoholism, etc.)
* Significant medical illnesses (e.g., cancer, meningitis, chronic obstructive pulmonary disease, cardiovascular disease, etc.)
* Cerebrovascular risk factors (e.g., hypertension, diabetes, elevated cholesterol, etc.)
* Use of psychoactive medications (e.g., barbiturates, benzodiazepines, chloral hydrate, haloperidol, lithium, carbamazepine, phenytoin, citalopram, escitalopram, fluoxetine, diazepam, etc.)
* Smell or taste dysfunction
* History of severe allergies requiring hospitalization for treatment
* History of severe asthma requiring hospitalization for treatment
* Habitual smoking
* History of eating disorders (e.g., anorexia nervosa, bulimia nervosa, binge-eating disorder, etc.)
* Dieting or fasting
* History of sleep disorders (e.g., obstructive sleep apnea, narcolepsy, insomnia, etc.) Magnetic implants (e.g., shunts or stents, aneurysm clips, surgical clips, cochlear implants, metal bone/joint pins, plates and screws, eyelid spring or wires, etc.)
* Electronic implants (e.g., implanted cardiac defibrillator, cardiac pacemaker, deep brain/spinal cord or nerve stimulator, internal electrodes/wires, medication infusion devices, etc.)
* History of metal working without proper eye protection, or injury with metal shrapnel or metal slivers
* Left-handedness
* Claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-01-14 (Actual); Primary Completion 2022-05-19 (Actual); Study Completion 2022-05-19 (Actual)

PRIMARY OUTCOMES:
Behavior an olfactory perceptual decision-making task | Up to 24 hours after the intervention
  Food-like perceptual responses to binary food-nonfood odor mixtures

SECONDARY OUTCOMES:
Resting-state functional magnetic resonance imaging | Up to 24 hours after the intervention
  Resting-state activity determined by functional magnetic resonance imaging

CONTACTS AND LOCATIONS:
Overall Officials: Thorsten Kahnt, PhD, Principal Investigator — Associate Professor; Christina Zelano, PhD, Principal Investigator — Assistant Professor
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Data underlying published results may be shared
Time Frame: Data may be shared upon publication
Access Criteria: Data can be obtained from the PI for non-profit purposes upon reasonable request